CLINICAL TRIAL: NCT01603836
Title: Allograft Alone Versus Allograft With Bone Marrow Concentrate for the Healing of the Instrumented Posterolateral Lumbar Fusion
Brief Title: Study Confirms or Refutes the Hypothesis That the Autologous Bone Marrow Concentrate Together With the Allograft is a Better Alternative for the Posterolateral Fusion in Spine Surgery Than the Allograft Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Znojmo (Other)
Responsible Party: Principal Investigator, Komzak Martin, M.D., Principal Investigator, Hospital Znojmo
Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PLFBMC
Record Dates: First submitted 2012-05-15; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Spondyloarthrosis, Spondylosis
Keywords: Lumbar spine; Posterolateral fusion; Allograft; Bone marrow concentrate; Mesenchymal stem cells; Fusion rate
MeSH Terms: conditions — Spondylarthritis; Spondylosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- bone marrow concentrate (Experimental): In forty cases, the posterolateral fusion was done with spongious allograft chips alone (Group I). In another forty cases, spongious allograft chips were mixed with BMC (Group II), where the mesenchymal stem cell (MSCs) concentration was 1.74 x104/L at average (range, 1.06-1.98 x104/L). Patients were scheduled for anteroposterior and lateral radiographs at 12 and 24 months after the surgery and for CT scanning at 24 months after the surgery. Fusion status and the degree of mineralization of the fusion mass were evaluated separately by two radiologists blinded to patient group affiliation.
  Interventions: Biological: bone allogaft with bone marrow concentrate

INTERVENTIONS:
Biological: bone allogaft with bone marrow concentrate — In forty cases, the PLF was done with spongious allograft chips alone (Group I). In another forty cases, spongious allograft chips were mixed with BMC (Group II), where the mesenchymal stem cell (MSCs) concentration was 1.74 x104/L at average (range, 1.06-1.98 x104/L). Patients were scheduled for anteroposterior and lateral radiographs at 12 and 24 months after the surgery and for CT scanning at 24 months after the surgery. Fusion status and the degree of mineralization of the fusion mass were evaluated separately by two radiologists blinded to patient group affiliation.

SUMMARY:
The use of autologous mesenchymal stem cell (MSCs) in form of the BMC in combination with allograft is an effective option how to enhance the Posterolateral Fusion (PLF) healing. Allograft by itself is not an effective material as a posterior onlay graft for the PLF in adult surgery.

DETAILED DESCRIPTION:
The study was prospective, randomized, controlled and blinded. Eighty patients with degenerative disease of the lumbar spine underwent instrumented lumbar or lumbosacral PLF. In forty cases, the PLF was done with spongious allograft chips alone (Group I). In another forty cases, spongious allograft chips were mixed with BMC (Group II), where the mesenchymal stem cell (MSCs) concentration was 1.74 x104/L at average (range, 1.06-1.98 x104/L). Patients were scheduled for anteroposterior and lateral radiographs at 12 and 24 months after the surgery and for CT scanning at 24 months after the surgery. Fusion status and the degree of mineralization of the fusion mass were evaluated separately by two radiologists blinded to patient group affiliation.

ELIGIBILITY:
Inclusion Criteria:

* degenerative disc disease or degenerative spondylolisthesis

Exclusion Criteria:

* vertebral fractures,
* infections or spinal neoplasms,
* non-rigid instrumentations,
* medication affecting bone mineralization (e.g., corticosteroids),
* body mass index higher than 35,
* systemic diseases,
* blood disease and/or immunosuppressant treatment and/or dicoumarol therapy;
* immunosuppressant and/or neoplastic and/or infectious diseases.

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The improvement of the fusion of the posterolateral fusion measured on X-rays | 12 months after the surgery
  Patients were scheduled for anteroposterior and lateral radiographs at 12 and 24 months after the surgery and for CT scanning at 24 months after the surgery. Fusion status and the degree of mineralization of the fusion mass were evaluated separately by two radiologists blinded to patient group affiliation.
The improvement of the fusion of the posterolateral fusion measured on X-rays and CT scans. | 24months after the surgery
  Patients were scheduled for anteroposterior and lateral radiographs at 12 and 24 months after the surgery and for CT scanning at 24 months after the surgery. Fusion status and the degree of mineralization of the fusion mass were evaluated separately by two radiologists blinded to patient group affiliation.